CLINICAL TRIAL: NCT02235597
Title: Improving Healthcare Systems for Access to Care by Underserved Patients
Acronym: PCORI
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Arizona State University (Other); Parkview Health (Other)
Responsible Party: Principal Investigator, Huanmei Wu, Associate Professor BioHealth Informatics, Indiana University
Other Study IDs: PCORI-WU-4198014; Improving Healthcare Systems (Other Grant/Funding Number: IH -12-11-5488)
Record Dates: First submitted 2014-09-03; First posted 2014-09-10 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Health Services Accessibility
Keywords: patient access; patient centered care; scheduling; access barriers; improve efficiency; decision making tools; underserved

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients and Staff of Community Clinics: Patients and Staff of Community Clinics who shared strategies and solutions to overcome barriers to accessing health care

SUMMARY:
The investigators seek to improve health systems so underserved people, patients without insurance, Medicaid, Medicare, as well as self pay and their caregivers can better access health care for common problems and acute care needs (same day appointments).

DETAILED DESCRIPTION:
There are different types of participants in this study. Measurements will be assessed with a questionnaire. The first category includes patients, caregivers, clinical and operational leaders, and researchers who will be invited for the Delphi study to identify potential barriers to access and strategies to improve access. The second category includes clinic staff (physicians, nurses, medical assistants, registrars, etc.) and patients who will be interviewed during their clinic visits to identify key processes and patients' opinion about barriers to access. The third category includes all enrolled patients to identify the patient population characteristics. The fourth category includes the patients and providers of CHCs in the participating clinics who will be surveyed to assess experience with access to care and satisfaction with the changes in workflow and efficiency.Category 1: Delphi study. The investigators will invite 50-60 individuals (patients, caregivers, clinical and operational leaders, and researchers) for a panel size of 40-50. Category 2: Key Informant Interviews (Patients and clinic staff (physicians, nurses, medical assistants, registrars, etc). The investigators will interview at least one patient every time we go to the participating clinics. The investigators plan to visit each of the participating CHCs approximately every two months. The investigators expect to interview approximately 12 patients at each clinic each year, for a total of 84 each year at the seven clinics. Thus, the total number of patients interviewed will be 252 in three years (12 patients / clinic x 7 clinics = 84 patients per year). The interview questions will be related to access barriers and efficiency of clinic processes. The investigators will receive the consent of the patient before starting the interview. The investigators will use IRB-approved consent forms for the study. The investigators will interview ten staff members during each visit to identify the key processes. The investigators anticipate interviewing approximately 8 providers and staff in each clinic during our bimonthly visits, as well as 3-4 during our bimonthly phone calls during the project period. This is expected to total 12 staff (including providers and managers) every two months at each clinic, or 6 x 12 = 72. This should total 72 x 7 = 504 at all the clinics each year. Some of these interviews will be quite brief, lasting only a few minutes, while others may last 45-60 minutes. Category 3: The investigators will collect de-identified patient data for the patient populations cared for by the participating CHCs, that will include age, gender, race, marital status, education, language, income, insurance, distance to healthcare facility, reason of the visit, diagnoses, co-morbidities, number of regular visits, visit types and durations, provider types, and time between visits. The investigators will work with IT and/or quality improvement staff at each of the CHCs to develop standard procedures to retrieve and de identify the data from electronic medical records and scheduling system. The investigators will analyze the data to determine patient population characteristics and care needs to inform the simulation models and analysis of impact of the interventions. In 2011, the total number of patients seen in seven partner clinic systems were approximately 130,000. However, the partner clinics provide care services at several sites. The investigators will choose a single site from each CHC system and analyze the data for the patients who had at least two prior visits to the selected site within two years prior to baseline. The investigators expect to analyze the visits for 60,000 patients. The data for each clinic will be analyzed separately. Category 4; The investigators anticipate surveying a sample of patients at each of the clinics to assess familiarity with how to obtain access to care, knowledge of the intervention and satisfaction with access. This will be a blinded (deidentified survey) and not linked to any individual data, other than study site. The investigators anticipate sampling 100 patients at each site, including approximately 65 patients who participate at each site., per site. In this study, the investigators will not consider special vulnerable populations (fetuses, neonates, prisoners, and institutionalized individuals).

ELIGIBILITY:
Inclusion Criteria:

* patient at an approved site Community health clinic and over 18 yrs of age.

Exclusion Criteria:

* do not receive care at an approved site Community health clinic and/or under 18 yrs of age.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community Clinic patient Population
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
patients will have improved access to providers | 2 years
  Patients in participating clinics will report improved access to providers for acute and regularly occurring appointments

CONTACTS AND LOCATIONS:
Overall Officials: Huanmei Wu, PhD, Principal Investigator — Indiana University
Locations (7):
- United States (7):
  - Valley Professionals Community Health Center, Cayuga, Indiana
  - North Central Nursing Clinics, Delphi, Indiana
  - Shalom Health Center, Indianapolis, Indiana
  - HealthNet Health Center, Indianapolis, Indiana
  - Riggs Community Health Center, Lafayette, Indiana
  - Open Door Community Health Clinic, Muncie, Indiana
  - North Shore Health Center, Portage, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Coulter A, Locock L, Ziebland S, Calabrese J. Collecting data on patient experience is not enough: they must be used to improve care. BMJ. 2014 Mar 26;348:g2225. doi: 10.1136/bmj.g2225. No abstract available. PMID 24671966
- [Result] Carman KL, Dardess P, Maurer M, Sofaer S, Adams K, Bechtel C, Sweeney J. Patient and family engagement: a framework for understanding the elements and developing interventions and policies. Health Aff (Millwood). 2013 Feb;32(2):223-31. doi: 10.1377/hlthaff.2012.1133. PMID 23381514